CLINICAL TRIAL: NCT03308656
Title: Uterocervical Angle in Success of Induction of Labor
Brief Title: Uterocervical Angle in Induction of Labor
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, MD, Director of labor room, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2017/239
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Labor Induction, Third Trimester
Keywords: uterocervical angle, labor induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Induced labor in term pregnancies: 100 singleton nulliparous patients are planning to complete the study period. Study group constitute of third trimester pregnancies between 37-40 weeks of gestation. All participants were nulliparous and had no systemic illnesses. The uterocervical angle will be measured in all participants before the induction of labor.
  Interventions: Other: uterocervical angle

INTERVENTIONS:
Other: uterocervical angle — uterocervical angle is the angle between lower segment of uterus and cervix

SUMMARY:
To evaluate the performance of uterocervical angle (UCA) in the prediction of labor induction.

DETAILED DESCRIPTION:
Induction of labor is a common procedure in obstetrics. In recent years, uterocervical angle (UCA) emerged as a new ultrasound parameter in the prediction of labor. Dziadosz et al concluded that the performance of UCA was even better than the cervical length in their cohort. A wide UCA during second trimester shown to have an increased risk of preterm labor and narrow angle was less likely to have labor.

The investigators are aimed to investigate predictive role of both cervical length and UCA in the labor induction in third trimester of pregnancy.The investigators focused on nulliparous women who are taking dinoproston for the cervical preparation and aim to measure their UCA.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous singleton pregnancy
* no previous systemic illnesses

Exclusion Criteria:

* abnormal Pap smear
* previous cesarean section
* history of dilatation and curettage (D&C)
* history of LEEP and cervical conization

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant population undergoing labor induction in the third trimester
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
uterocervical angle | once at the beginning of enrollment
  the angle between the lower segment of uterus and cervix

CONTACTS AND LOCATIONS:
Overall Officials: Alev Aydin, MD,ObGyn, Study Director — Kanuni SSTRH
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Uterocervical angle: a novel ultrasound screening tool to predict spontaneous preterm birth. — http://www.ncbi.nlm.nih.gov/pubmed/27018466